CLINICAL TRIAL: NCT03746457
Title: Alcohol and ART Adherence: Assessment, Intervention and Modeling in India
Brief Title: Alcohol and ART Adherence in India
Acronym: RISHTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Institute for Community Research (Unknown); International Center for Research on Women (Unknown); Population Council (Other)
Responsible Party: Principal Investigator, Stephen Schensul, Professor, UConn Health
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: U01AA021990 (NIH)
Record Dates: First submitted 2018-11-11; First posted 2018-11-19 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Alcohol Consumption; HIV Infection Primary
MeSH Terms: conditions — Alcohol Drinking | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Participants in the three experimental ART Centers received three cycles of intervention, while two ART Centers served as the controls. In the first cycle, participants in the three experimental Centers each received individual counseling, group intervention (GI) and collective advocacy (CA). In Cycle 2, participants in each experimental center received a second intervention (e.g. GI + CA) and in the third cycle, participants in each experimental Center received a third intervention (GI + CA + IC). In addition, in Cycle 3, the participants in one of the Control Centers received an integrated package of IC-GI-CI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control ART Center (No Intervention): Control arm with no intervention throughout the course of the study
- Control and Cycle 3 integrated package (Active Comparator): Control arm in Cycles 1 and 2 and in Cycle three converts to experimental
  Interventions: Behavioral: Behavioral intervention
- GI + CA + IC (Experimental): Receives one alternative sequence of three interventions
  Interventions: Behavioral: Behavioral intervention
- IC + GI + CA (Experimental): Receives a second alternative sequence of three interventions
  Interventions: Behavioral: Behavioral intervention
- CA + IC + GI (Experimental): Receives a third alternative sequence of three interventions
  Interventions: Behavioral: Behavioral intervention

INTERVENTIONS:
Behavioral: Behavioral intervention — Individual counseling, group intervention, collective advocacy
  Arms: CA + IC + GI; Control and Cycle 3 integrated package; GI + CA + IC; IC + GI + CA

SUMMARY:
The focus of this project was to reduce alcohol consumption among male "persons living with HIV" (PLHIV) on antiretroviral treatment (ART) at government hospitals in urban Maharashtra, India and factors associated with both these outcomes including depression, stigma, social support networks, quality of life and health status. The project consisted of three phases; formative research, implementation of multilevel interventions and analysis of process and outcome data. The project utilized a crossover design to compare outcomes of individual interventions and the sequences of intervention.

DETAILED DESCRIPTION:
The focus of this project was to reduce alcohol consumption among male "persons living with HIV" (PLHIV) on antiretroviral treatment (ART) at government hospitals in urban Maharashtra, India and factors associated with both these outcomes including depression, stigma, social support networks, quality of life and health status.

The project consisted of three phases; formative research, intervention implementation and analysis and dissemination. Formative research included key informant interviews and observation at the ART Centers, screening of close to 10,000 patients to identify male PLHIV who met the eligibility criteria, a baseline survey instrument (T1) that assessed a wide range of variables associated with the outcome variables and modeling alternative intervention programs for impact and cost effectiveness. Of 13 ART Centers in the Mumbai, Navi Mumbai, and Thane areas of Maharashtra, five ART Centers were selected for the project with a sample of 940 male PLHIV, 188 from each of the five ART Centers.

The second phase of the project was the development and implementation of three interventions assigned randomly to each of the experimental ART Centers with two of the Centers selected randomly as controls. The interventions were individual counseling (IC), group intervention (GI) and collective advocacy (CA). In Cycle 1 of the intervention phase, the interventions were implemented in each of three experimental ART Centers. In Cycle 2, each of the experimental centers received a second intervention (e.g. GI in Cycle 1+ IC in Cycle 2) and in Cycle 3 each of the experimental Centers received the third intervention (GI in Cycle 1 + IC in Cycle 2 + CA in Cycle 3). In addition, in Cycle 3, one of the two controls received an integrated package of IC, GI and CA. This crossover design test the sequencing and packaging of multi-level interventions for behavior change by examining the efficacy of any one intervention versus control, any two combinations of interventions versus controle, all interventions versus control and the integrated package versus control.

The IC intervention involved one-on-one interaction with a project counselor involving a pre-intervention session in which the PLHIV participant selected the priority issues to be discussed and four additional sessions to address tensions and anxieties, stigma and disclosure, relationships and alcohol and adherence. The sessions were facilitated by in the use of a tablet both to structure the interaction and to collect process data. GI involved four sessions in which 6-10 PLHIV were gathered for intervention on healthy living with HIV, tension, relationships and alcohol and adherence. CA involved groups of 10-15 PLHIV in five sessions in which the focus was on increasing the capacity of participants to advocate both for themselves and a collective group for issues that affected PLHIV human rights, entitlements and services.

The third and current phase of the project is analysis of qualitative data including key informant and in-depth interviews with PLHIV and assessments of fidelity and acceptability of the interventions and quantitative data that includes the screening instrument and baseline (T1) and follow-up outcome data (T2, T3, T4 follow-up surveys after each intervention for both experimental and control centers. This phase will also involve dissemination of results to the National AIDS Control Organizations and its subsidiaries at the State and District levels, the participating ART Centers and to Positive Peoples' Networks at the state and national levels and to national and international meetings and publications.

ELIGIBILITY:
Inclusion Criteria:

* Male
* age 18-60
* six months or more on ART
* consumed alcohol at least once in the last 30 days

Exclusion Criteria:

* Female
* outside the age range
* less than 6 months on ART
* did not consume alcohol in the last 30 days

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Based on self-representation
Enrollment: 940 (Actual)
Dates: Start 2015-05-10 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Measurements to assess change made at four (4) time points; baseline and 80-120 days post intervention for each of three cycles of intervention, approximately 9 months apart.
  Alcohol problem drinking measured by 10-item Alcohol Use Disorders Identification Test (AUDIT) developed by WHO and validated in India. The responses for each item were scored from 0 to 4. The total score range from 1 to 32 with higher scores indicating a high level of alcohol use. The total scores categorized as low risk (0-7), moderate risk (8-15), high risk (≥ 16).
The AIDS Clinical Trials Group (ACTG) Adherence Questionnaire | Measurements to assess change made at four (4) time points; baseline and 80-120 days post intervention for each of three cycles of intervention, approximately 9 months apart.
  The AIDS Clinical Trials Group (ACTG) Adherence Questionnaire, 4-day recall, involves a self-report of the number of times an HIV+ individuals have taken their ART medication in relation to the number of times prescribed, for the previous four (4) day period. if the prescription is twice per day, then a single missed dose results in a score of 1/8 or 12.5%.
CD-4 count | Measurements to assess change made at four (4) time points; baseline and 80-120 days post intervention for each of three cycles of intervention, approximately 9 months apart.
  The CD4 count measures the functioning of the immune system the number of white blood (T) cells that fight infection. As HIV infection progresses, the number of these cells declines.
Viral Load | Measurements to assess change made at four (4) time points; baseline and 80-120 days post intervention for each of three cycles of intervention, approximately 9 months apart.
  The HIV viral load test is used to determine the level of HIV infection in a person diagnosed with the disease. HIV viral load testing measures the amount of HIV genetic material (RNA) in the blood and reports how many copies per ml of the virus are present

SECONDARY OUTCOMES:
Center for Epidemiologic Studies-Depression scale (CES-D) | Measurements to assess change made at four (4) time points; baseline and 80-120 days post intervention for each of three cycles of intervention, approximately 9 months apart.
  Depressive symptoms are measured using the 10-item Center for Epidemiologic Studies-Depression (CES-D) scale which covers depressed mood, feelings of guilt, worthlessness, and helplessness, loss of appetite, and sleep disturbance, and has been validated in India. The total score ranges from 0 to 30. The resulting scale was skewed, so it was transformed to a categorized variable by using the standardized cut of of 10 to distinguish none/mild (0-9) from moderate (10-14) and severe (15 or higher) depressive symptoms.
HIV Internalized Stigma | Measurements to assess change made at four (4) time points; baseline and 80-120 days post intervention for each of three cycles of intervention, approximately 9 months apart.
  HIV-related self stigma 16-item scale measuring rejection by family, friends, workplace and services, derived from Berger's HIV stigma scale validated in India that covers three domains: fears related to disclosure (6 items); negative self-image (5 items); and concerns with public attitudes about people with HIV (5 items). Participants responded to each question using a four-item Likert scale (strongly disagree = 1, disagree = 2, agree = 3 and strongly agree = 4). The total score ranged from 16-64 with higher scores indicating greater perception of HIV related self-stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Schensul, PhD, Principal Investigator — UConn Health; Jean J Schensul, PhD, Principal Investigator — Institute for Community Research; Niranjan Saggurti, PhD, Principal Investigator — Population Council, India Country office; Avina Sarna, MD, Principal Investigator — Population Council, India Country office
Locations (1):
- University of Connecticut Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be available in a de-identified status, three years after termination of the project
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: February 1, 2023
Access Criteria: All researchers in research organizations

REFERENCES:
- [Result] Schensul SL, Ha T, Schensul JJ, Vaz M, Singh R, Burleson JA, Bryant K. The Role of Alcohol on Antiretroviral Therapy Adherence Among Persons Living With HIV in Urban India. J Stud Alcohol Drugs. 2017 Sep;78(5):716-724. doi: 10.15288/jsad.2017.78.716. PMID 28930059
- [Result] Schensul JJ, Ha T, Schensul S, Sarna A, Bryant K. Identifying the Intersection of Alcohol, Adherence and Sex in HIV Positive Men on ART Treatment in India Using an Adapted Timeline Followback Procedure. AIDS Behav. 2017 Nov;21(Suppl 2):228-242. doi: 10.1007/s10461-017-1916-1. PMID 28993911
- [Result] Ruggles KV, Patel AR, Schensul S, Schensul J, Nucifora K, Zhou Q, Bryant K, Braithwaite RS. Betting on the fastest horse: Using computer simulation to design a combination HIV intervention for future projects in Maharashtra, India. PLoS One. 2017 Sep 5;12(9):e0184179. doi: 10.1371/journal.pone.0184179. eCollection 2017. PMID 28873452
- [Result] Patel AR, Ruggles KV, Nucifora K, Zhou Q, Schensul S, Schensul J, Bryant K, Braithwaite RS. Evaluating Alternative Designs of a Multilevel HIV Intervention in Maharashtra, India: The Impact of Stakeholder Constraints. MDM Policy Pract. 2018 Oct 16;3(2):2381468318803940. doi: 10.1177/2381468318803940. eCollection 2018 Jul-Dec. PMID 30349875
- [Derived] Ha T, Pham TQ, Misra S, Su TW, Ha L, Cunningham SD, Carandang RR, Schensul SL. Impact of multilevel interventions on reducing reasons for drinking among men living with HIV. AIDS Care. 2025 Oct;37(10):1696-1705. doi: 10.1080/09540121.2025.2547030. Epub 2025 Aug 22. PMID 40844326
- [Derived] Ha T, Shi H, Pham BN, Dsouza A, Shrestha R, Kuchipudi SV, Luu HN, Le NT, Schensul SL. Assessing the Effectiveness of Multilevel Intervention Sequences on "Tension" Among Men Living with HIV: A Randomized-Control Trial. Int J Behav Med. 2025 Oct;32(5):647-657. doi: 10.1007/s12529-024-10310-5. Epub 2024 Jul 29. PMID 39073518
- [Derived] Ha T, Shi H, Shrestha R, Gaikwad SS, Joshi K, Padiyar R, Schensul SL. The Mediating Effect of Changes in Depression Symptoms on the Relationship between Health-Related Quality of Life and Alcohol Consumption: Findings from a Longitudinal Study among Men Living with HIV in India. Int J Environ Res Public Health. 2023 Apr 18;20(8):5567. doi: 10.3390/ijerph20085567. PMID 37107849
- [Derived] Schensul SL, Ha T, Schensul JJ, Grady J, Burleson JA, Gaikwad S, Joshi K, Malye R, Sarna A. Multilevel and Multifactorial Interventions to Reduce Alcohol Consumption and Improve ART Adherence and Related Factors Among HIV Positive Men in Mumbai, India. AIDS Behav. 2021 Dec;25(Suppl 3):290-301. doi: 10.1007/s10461-021-03303-y. Epub 2021 May 20. PMID 34014429